CLINICAL TRIAL: NCT03858907
Title: Risk of Cytomegalovirus Disease or High Viremia in Seropositive Kidney Transplant Recipients Stratified by Quantiferon-CMV
Brief Title: Cytomegalovirus Risk in Seropositive Kidney Transplant Recipients Stratified by Quantiferon-CMV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: quantiferon-cmv_ktx
Record Dates: First submitted 2019-02-21; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Cytomegalovirus Infections; CMV; Kidney Transplant Infection
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
To evaluate the Quantiferon-CMV test ability to predict occurrence of cytomegalovirus (CMV) disease o treated infection after kidney transplantation. Patients studied are those already infected by CMV before transplantation ("seropositive"). Patients given thymoglobulin as induction therapy receive CMV prophylaxis with valganciclovir, while those given basiliximab undergo weekly monitoring for CMV viremia with preemptive treatment as needed.

DETAILED DESCRIPTION:
This study evaluates Quantiferon-CMV assay ability for CMV (cytomegalovirus) risk prediction in kidney transplant recipients. Quantiferon-Monitor ability to predict infection or graft rejection will be evaluated as an exploratory objective.

It is a prospective cohort study. The assumption is that CMV disease or preemptively treated viremia (dependent variable) may be predicted by Quantiferon-CMV result (independent variable). Quantiferon-CMV results will be masked for the assistant physician.

Patients are evaluated for eligibility on their hospital admission for kidney transplantation. Type of induction therapy follows current local protocol: thymoglobulin is given to sensitized patients against HLA - human leukocyte antigen (that is, PRA > 0%), and basiliximab to unsensitized patients (PRA = 0%). Initial maintenance immunosuppression includes prednisone, tacrolimus and mycophenolate sodium to all patients. If a patient is enrolled in the study, blood is drawn before transplantation for pre-transplant Quantiferon assays (CMV and Monitor).

For CMV disease prevention, transplant recipients undergo until day 90 post-transplant: either weekly CMV monitoring (qPCR - quantitative polymerase chain reaction - and pp65 antigenemia) and preemptive treatment if given basiliximab or antiviral prophylaxis if given thymoglobulin for induction. Cutoff values for preemptive treatment are 4,000 IU/ml of plasma for Abbott Real Time PCR or ≥ 4 cells/300.000 neutrophils for pp65 Antigenemia. After day 90 post-transplant, all participants undergo biweekly CMV monitoring until day 180 with preemptive treatment as needed.

Quantiferon-CMV results from 2 or 3 different moments (pre-transplant, day 30 and for patients given thymoglobulin also day 90) will be analyzed with subsequent occurrence of CMV disease/treated viremia. Analysis will be stratified by type of induction therapy. A high negative predictive value of pre-transplant or day 30 Quantiferon-CMV could indicate unneeded monitoring for preemptive treatment. On the other hand, a high positive predictive value for CMV occurrence could indicate the necessity of antiviral prophylaxis implementation.

Patients given thymoglobulin will undergo a third Quantiferon-CMV on day 90, at the end of their antiviral prophylaxis. This third Quantiferon-CMV may predict occurrence of late disease, together with clinical variables (low kidney graft function / glomerular filtration rate, lymphopenia or type of donor). A high positive predictive value for CMV disease/treated viremia could indicate the need for antiviral extension beyond 3 months.

Clinical and laboratory parameters evaluated also include: demographic and pre-transplant clinical data, monthly creatinine and blood cell counts, complement 3 fraction, total IgG, blood BK and EBV virus qPCR, CD4/CD8 cells counts, CMV serology, acute rejection and type of treatment, opportunistic and bacterial infections, post-transplant diabetes, maintenance immunosuppression, diabetes, delayed graft-function.

Multivariable logistic regression models will be tested for their performance to predict CMV disease/treated infection.

For the cost-effectiveness analysis, current strategy without QF-CMV will be compared with a simulated strategy with a QF-CMV-oriented CMV prevention. For this analysis, costs will be in the perspective of Hospital das Clinicas de Sao Paulo with values obtained part from micro-costing and part from secondary data.

ELIGIBILITY:
Inclusion Criteria:

* CMV IgG seropositivity before kidney transplant
* to provide signed Informed Consent

Exclusion Criteria:

* death or graft failure before day 19 post-transplant
* allergy to valganciclovir ou ganciclovir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients from a big tertiary hospital in Sao Paulo, Brazil
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2018-08-05 (Actual); Primary Completion 2020-08-05 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
CMV disease/treated infection occurrence according to Quantiferon-CMV result | 365 days
  To evaluate if QF-CMV (either pre or post-transplant) predicts occurrence of CMV disease or treated infection in CMV seropositive kidney recipients, stratified by type of induction therapy

SECONDARY OUTCOMES:
QF-CMV cutoff values | 365 days
  To define cut-off values of IFN-gamma production by Quantiferon-CMV that best predict CMV (disease or treated viremia) occurrence
CMV risk prediction index | 365 days
  To define the best predictive model for the occurrence of CMV, which includes QF-CMV and clinical/laboratory variables (donor type, kidney function and lymphocyte counts).
Association of CMV with clinical events | 365 days
  To evaluate the association of CMV infection with occurrence: acute rejection, bacterial or opportunistic infection and neutropenia
Association of CMV and patient and graft survivals | 365 days
  To analyze patient and graft survival stratified by CMV infection (Kaplan-Meier method)
Association of CMV and total IgG levels | 365 days
  To evaluate the association of CMV infection with serum IgG (immunoglobulin G) levels at 0, 1, 3, and 6 months post-transplant
Association of CMV and lymphocytes counts | 365 days
  To evaluate the association of CMV infection with blood CD4 and CD8 lymphocytes counts at 0, 1, 3, and 6 months post-transplant
Association of CMV and graft function | 365 days
  To evaluate the association of CMV infection with estimated glomerular filtration rate by Modification of Diet in Renal Disease formula (creatinine based) at 0, 1, 3, and 6 months post-transplant

OTHER OUTCOMES:
Infection and acute rejection prediction with Quantiferon-Monitor | 365 days
  To evaluate the discriminative ability of QF-Monitor results (in IU of interferon/ml) to predict occurrence of first acute rejection episode or any bacterial/opportunistic infection

CONTACTS AND LOCATIONS:
Overall Officials: Elias David-Neto, MD, PhD, Principal Investigator — Instituto do Coracao
Locations (1):
- Hospital das Clinicas, University of Sao Paulo School of MedicinE, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reusing JO Jr, Feitosa EB, Agena F, Pierrotti LC, Azevedo LSF, Kotton CN, David-Neto E. Cytomegalovirus prophylaxis in seropositive renal transplant recipients receiving thymoglobulin induction therapy: Outcome and risk factors for late CMV disease. Transpl Infect Dis. 2018 Oct;20(5):e12929. doi: 10.1111/tid.12929. Epub 2018 Jul 2. PMID 29809309
- [Background] Kotton CN, Kumar D, Caliendo AM, Huprikar S, Chou S, Danziger-Isakov L, Humar A; The Transplantation Society International CMV Consensus Group. The Third International Consensus Guidelines on the Management of Cytomegalovirus in Solid-organ Transplantation. Transplantation. 2018 Jun;102(6):900-931. doi: 10.1097/TP.0000000000002191. PMID 29596116
- [Background] David-Neto E, Triboni AH, Paula FJ, Vilas Boas LS, Machado CM, Agena F, Latif AZ, Alencar CS, Pierrotti LC, Nahas WC, Caiaffa-Filho HH, Pannuti CS. A double-blinded, prospective study to define antigenemia and quantitative real-time polymerase chain reaction cutoffs to start preemptive therapy in low-risk, seropositive, renal transplanted recipients. Transplantation. 2014 Nov 27;98(10):1077-81. doi: 10.1097/TP.0000000000000189. PMID 24839894
- [Background] Lisboa LF, Kumar D, Wilson LE, Humar A. Clinical utility of cytomegalovirus cell-mediated immunity in transplant recipients with cytomegalovirus viremia. Transplantation. 2012 Jan 27;93(2):195-200. doi: 10.1097/TP.0b013e31823c1cd4. PMID 22179399
- [Background] Fernandez-Ruiz M, Gimenez E, Vinuesa V, Ruiz-Merlo T, Parra P, Amat P, Montejo M, Paez-Vega A, Cantisan S, Torre-Cisneros J, Fortun J, Andres A, San Juan R, Lopez-Medrano F, Navarro D, Aguado JM; Group for Study of Infection in Transplantation of the Spanish Society of Infectious Diseases and Clinical Microbiology (GESITRA-SEIMC) and the Spanish Network for Research in Infectious Diseases (REIPI). Regular monitoring of cytomegalovirus-specific cell-mediated immunity in intermediate-risk kidney transplant recipients: predictive value of the immediate post-transplant assessment. Clin Microbiol Infect. 2019 Mar;25(3):381.e1-381.e10. doi: 10.1016/j.cmi.2018.05.010. Epub 2018 May 25. PMID 29803844
- [Background] Cantisan S, Lara R, Montejo M, Redel J, Rodriguez-Benot A, Gutierrez-Aroca J, Gonzalez-Padilla M, Bueno L, Rivero A, Solana R, Torre-Cisneros J. Pretransplant interferon-gamma secretion by CMV-specific CD8+ T cells informs the risk of CMV replication after transplantation. Am J Transplant. 2013 Mar;13(3):738-45. doi: 10.1111/ajt.12049. Epub 2013 Jan 11. PMID 23311355
- [Derived] Gibson L. An Interferon-gamma Release Assay for Evaluation of Cell-mediated Immunity in Infants With Congenital Cytomegalovirus Infection. Clin Infect Dis. 2021 Aug 2;73(3):374-375. doi: 10.1093/cid/ciaa700. No abstract available. PMID 32504089